CLINICAL TRIAL: NCT00438893
Title: The Long-Term Effect of Viscous Fibers, Soy Protein, and Plant Sterol Foods in Combination on Serum Cholesterol and Other Risk Factors for Cardiovascular Disease
Brief Title: Effects of a Long Term Dietary Portfolio and of Sequential Removal of Food Components From the Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canada Research Chairs Endowment of the Federal Government of Canada (Other Government); Natural Sciences and Engineering Research Council, Canada (Other); Loblaw Companies Limited (Industry); Almond Board of California (Other); Unilever R&D (Industry)
Responsible Party: Principal Investigator, David Jenkins, Principle Investigator, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB 03-043; HC-CT#100934
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Hyperlipidemia; Cardiovascular Diseases; Hypercholesterolemia
Keywords: Viscous dietary fiber; Soy protein; Nuts; Plant sterols; Dietary Portfolio; Compliance; Blood lipids; Blood pressure
MeSH Terms: conditions — Hyperlipidemias; Cardiovascular Diseases; Hypercholesterolemia; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A portfolio of cholesterol-lowering foods (Other): Dietary advice to consume a dietary portfolio of cholesterol-lowering foods
  Interventions: Dietary Supplement: Dietary portfolio of cholesterol-lowering foods

INTERVENTIONS:
Dietary Supplement: Dietary portfolio of cholesterol-lowering foods — A plant based dietary portfolio providing plant sterols (1.0g/1000 kcal), soy protein (22.5g/1000 kcal, viscous fibers 10 g/1000 kcal and almonds 22.5g/1000 kcal)

SUMMARY:
The purpose of this study is to evaluate the long term effectiveness of the dietary portfolio, consisting of viscous fibers, soy products, nuts and plant sterols, as well as the effects of removing single food components from the dietary portfolio on cholesterol reduction and other cardiovascular risk factors.

DETAILED DESCRIPTION:
We have shown in 1-month metabolic studies that a dietary portfolio, consisting of soy products, viscous fibers, almonds and plant sterols in the form of margarine, can lower cholesterol to the same extent as first generation statins (cholesterol-lowering drugs). However, the long-term effectiveness of the dietary portfolio is not known. Furthermore, it is not known to what extent each of the food components contribute to the cholesterol reductions observed. We wish to therefore evaluate the long term effects of the dietary portfolio as well as the effects of removing single food components from the dietary portfolio on cholesterol reduction and other cardiovascular risk factors. We believe the removal of single food components will result in a reduction of the cholesterol-lowering effect to a similar extent as predicted with the cholesterol reductions observed when the food component is consumed alone.

Method:

66 subjects will be recruited for a 6-month to 5 year long-term dietary portfolio study with the option for continuation (re-consenting) at the end of 6, 12 or 24 months. The active dietary components consist of viscous fibers (including oat bran), soy products (including soy milk), almonds and plant sterols (sterol-enriched margarine). Lipids, blood pressure, body weight, and routine biochemical and hematology analyses will be performed over the 5 year period, with lipids and blood pressure measured at 2 monthly intervals. 40-50 subjects on the long term dietary portfolio study, all of whom will have been on the diet for at least 1 year, will be asked to remove a specific food component from their regular dietary portfolio for a 10 week period. After the 10 week period, subjects will be asked return to the normal dietary portfolio with all food components consumed and continue on the long-term dietary portfolio.

Bloods will be taken at weeks 0, 6 and 10 of the food component removal period; and at 2-monthly intervals for 20 weeks prior to and after the 10 week period while on the long-term dietary portfolio with all food components.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and postmenopausal women currently enrolled in the long-term portfolio study
* Body mass index <32 kg/m2
* Constant body weight over last 6 months preceding the onset of the study
* Fasting LDL-cholesterol concentration >4.1 mmol/L at diagnosis

Exclusion Criteria:

* women of child-bearing potential
* major cardiovascular event (stroke or myocardial infarction)
* positive molecular diagnosis of familial hypercholesterolemia
* secondary causes of hypercholesterolemia (hypothyroidism, unless treated & on a stable dose of L-thyroxine, renal or liver disease)
* use of cholesterol-lowering medications
* serum triglycerides >4.5 mmol/L
* blood pressure > 145/90 mmHg
* diabetes and/or major disorders such as liver disease, renal failure or cancer
* major surgery <6 months prior to randomization
* alcohol consumption >2 drinks per day

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2003-09-01 (Actual); Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Total cholesterol | At weeks 0, 2,4, 8,12, 18, 24, 34, 44, 52; then every 2 months to a total of 5 years
LDL cholesterol | At weeks 0, 2,4, 8,12, 18, 24, 34, 44, 52; then every 2 months to a total of 5 years
C-reactive protein | At weeks 0, 12, 24, 34, 52; then every 6 months to a total of 5 years
Blood pressure | At weeks 0, 2,4, 8,12, 18, 24, 34, 44, 52; then every 2 months to a total of 5 years

SECONDARY OUTCOMES:
Body Weight | At weeks 0, 2,4, 8,12, 18, 24, 34, 44, 52; then every 2 months to a total of 5 years
Apolipoprotein A1 and B | At weeks 0, 2,4, 8,12, 18, 24, 34, 44, 52; then every 2 months to a total of 5 years
Lp(a) | At weeks 0, 24, 52; then every 6 months to a total of 5 years
Routine Biochemistry and hematology measurements | At week 0, 12, 24 and every 6 months to 5 years
Compliance to dietary portfolio components | At years, 1, 2, 3, 4 and 5
24 hour urinary markers and electrolytes (optional) | At week 0 and end of years 1, 2, 3, 4 and 5
Oxidative stress markers | week 0 and every 6 months to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: David JA Jenkins, MD, PhD, DSc, Principal Investigator — Department of Nutritional Sciences, Faculty of Medicine, University of Toronto
Locations (1):
- Clinical Nutrition & Risk Factor Modification Centre, St. Michael's Hospital Health Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Jenkins DJ, Kendall CW, Faulkner D, Vidgen E, Trautwein EA, Parker TL, Marchie A, Koumbridis G, Lapsley KG, Josse RG, Leiter LA, Connelly PW. A dietary portfolio approach to cholesterol reduction: combined effects of plant sterols, vegetable proteins, and viscous fibers in hypercholesterolemia. Metabolism. 2002 Dec;51(12):1596-604. doi: 10.1053/meta.2002.35578. PMID 12489074
- [Background] Jenkins DJ, Kendall CW, Marchie A, Faulkner DA, Wong JM, de Souza R, Emam A, Parker TL, Vidgen E, Lapsley KG, Trautwein EA, Josse RG, Leiter LA, Connelly PW. Effects of a dietary portfolio of cholesterol-lowering foods vs lovastatin on serum lipids and C-reactive protein. JAMA. 2003 Jul 23;290(4):502-10. doi: 10.1001/jama.290.4.502. PMID 12876093
- [Background] Jenkins DJ, Kendall CW, Marchie A, Faulkner D, Vidgen E, Lapsley KG, Trautwein EA, Parker TL, Josse RG, Leiter LA, Connelly PW. The effect of combining plant sterols, soy protein, viscous fibers, and almonds in treating hypercholesterolemia. Metabolism. 2003 Nov;52(11):1478-83. doi: 10.1016/s0026-0495(03)00260-9. PMID 14624410
- [Result] Jenkins DJ, Kendall CW, Faulkner DA, Nguyen T, Kemp T, Marchie A, Wong JM, de Souza R, Emam A, Vidgen E, Trautwein EA, Lapsley KG, Holmes C, Josse RG, Leiter LA, Connelly PW, Singer W. Assessment of the longer-term effects of a dietary portfolio of cholesterol-lowering foods in hypercholesterolemia. Am J Clin Nutr. 2006 Mar;83(3):582-91. doi: 10.1093/ajcn.83.3.582. PMID 16522904
- [Derived] Jenkins DJ, Kendall CW, Nguyen TH, Marchie A, Faulkner DA, Ireland C, Josse AR, Vidgen E, Trautwein EA, Lapsley KG, Holmes C, Josse RG, Leiter LA, Connelly PW, Singer W. Effect of plant sterols in combination with other cholesterol-lowering foods. Metabolism. 2008 Jan;57(1):130-9. doi: 10.1016/j.metabol.2007.08.016. PMID 18078870